CLINICAL TRIAL: NCT06088576
Title: Using a Digital Mental Health Application in the Adolescent's Care Pathway.
Brief Title: Using a Digital Application for Adolescents in Dropout of Care in Mental Health : Facilitate the Return in Classic Care With Telepsychiatry, Tchats, Forums and a Home Medical Team.
Acronym: TOGETHER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dominique JANUEL (Other)
Responsible Party: Sponsor-Investigator, Dominique JANUEL, Head of clinical research unit, Centre hospitalier de Ville-Evrard, France
Organization: Centre hospitalier de Ville-Evrard, France (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A00722-41
Record Dates: First submitted 2022-07-20; First posted 2023-10-18 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Mental Health
Keywords: adolescent; digital mental health application; digital application; telepsychiatry; telemedecine
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The group consists of teenagers between 11 and 18 years old, recruited by professionals of medical-psychological center, Child Protection, school medicine college and high school as well as pediatric emergencies. The group will have access to the digital mental health application for 6 months. Assessments will take place at different times.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- test group (Other): Following the inclusion interview, adolescents has access to the Together application.
  During the duration of the support, he will have access to the news, chat and forum.
  Teenager have 8 working days to appropriate the application. For 1 month, the chat can be used without any other means of communication. A chat is limited to 20-30 minutes, after that, a teleconsultation can be offer. At the end of the 1 month, teleconsultations or a home visit are possible (30 to 45 minutes). They are done between 1 to 4 sessions in the month. Following the orientation, the psychologists take over the visio for the next 2 months, up to 2 to 4 interviews per month. Teleconsultation appointments are made on the calendar of the application by the professional after obtaining advice from teenagers.
  At the beginning of the 5th month of care, the professionals set up a mixed distance/presential care with the youth. They propose home visits, individual or group interviews on site.
  Interventions: Other: Together

INTERVENTIONS:
Other: Together — Tchat : limited to 20-30 minutes per day. With a member of the team Together. For teleconsultations : First teleconsultation, during the first month (1 to 4 sessions/month), are made by nurse and/or educator. After that, it is psychologists who do the teleconsultations (2 to 4 sessions/month). It's during 30 to 45 minutes.
  Home visits, individual or group interviews on site are possible after 4 month.

SUMMARY:
Clinical experience has shown that adolescents have great difficulties in getting to mental health care centers. The investigators want to find a specific way to follow up with the adolescent public. This study sets up a digital mental health application offering a tele-consultation space, a chat space with mental health professionals, a forum space, a news and therapeutic education space. The objective of the study is to evaluate the acceptance of the digital tool by the adolescent between 11 and 18 years old. To do this, the investigators determine the number of connections to the tool during the 6 months of support.

DETAILED DESCRIPTION:
The purpose of the CPP application is the creation of an innovative psychiatric device combining a digital application of mental health for adolescents with a mobile team, anchored within the I03 pole of the Public Health Establishment of Ville-Evrard.

This Together digital application includes a space for news, chat, peer-to-peer forum and video consultation. We propose an action-research protocol because this project was born of questions related to the terrain raising the problem of the difficulty of access to the care of adolescents in the territory of Pole 93I03.

Action research is aimed at adolescents aged 11 to 18, whose medical, paramedical and school partners have observed mental suffering (ill-being, inappropriate behaviour, dropping out of school) but who are not or no longer enrolled in mental care. It aims to use a digital application backed by a mobile team to improve access to the mental health care system for adolescents.

The research issue would be formalized in these terms: would the Together mental health application, combined with a mobile team, allow access to a path of care for the adolescent?

HYPOTHESIS We hypothesize that adolescents will accept the digital tool, using it regularly and that this will ultimately facilitate access to mental care.

OBJECTIVES The main objective of this study is to assess the acceptance of the digital tool by the young person. Acceptance here depends on the regular use of the Together app by the teenager. The secondary objectives are to assess the percentage of adolescents starting face-to-face management within sector structures; the percentage of adolescents observing a better-be, to observe the quality of the support via the dual device digital application/mobile team.

METHOD The action-research takes place over a year, with a panel of 50 teenagers. After a pre-inclusion interview by the partners to talk about the research-action device to the teenager, he is offered an inclusion interview informing him of the research, the consent and the use of the digital application. Different evaluations are then spent at different times of action research to evaluate the main objective and secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Aged 11 - 18 years old
* Observation of mental suffering (ill-being, inappropriate behaviour, dropping out of school) following a medical, psychological or educational interview in the school, medical, paramedical, personal setting by a practitioner trained for this type of observation.
* Have access to the Internet via smartphone and have a sufficient mastery of the tool (spoken and read French).
* First-time arrivals on the sector who does not want management or dropout of care.
* Not to be or no longer to be followed therapeutically by a psychologist or psychiatrist in the liberal or inter-sector.
* Informed consent of the patient.

Exclusion Criteria:

* Disabling Motor Disorders (Cerebral Motor Disability).
* Heavy deficiency.
* Infant psychosis with strong relationship problems. .
* Withdrawal of care without degradation of the psychic state. .
* Is not in the pole 93I03 ( EPS Ville-Evrard).

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The number of connections to the application during the 6 months of support. | Day 0 to Month 6
  The data tool will collect and count the number of connections on the application, the number of chat, video, phone call and like given to the news. The software CORTEXTE (digital patient record), will count the number of acts performed with the young person.
The quality of the interaction between the user and the application assessed by AttrakDiff 2. | Month 3 and Month 6
  The Investigators use AttrakDiff 2, a validated self-assessment scale (Hassenzahl, Burmester and Kollet, 2003). It is consists in 28 items. Each item has 2 contrasting words (semantic differentiators), separated by a 7-point scale. The scale is divided into 7 pairs of words evaluating respectively: pragmatic aspects, the overall attractiveness of the interactive system, hedonic aspects - divided into two subscales: identification and stimulation. The purpose of this measure is to assess the global quality of the interaction between the user and the application.

SECONDARY OUTCOMES:
Behavioral disorders assessed by the score of Strengths and Difficulties Questionnaire(SDQ). | Day 0, month 3, month 6, month 12
  The self-administered questionnaire, validate by Goodman, 2015, for adolescents aged 11 to 16 consists of 25 questions to assess behavioral and adjustment problems in 5 main areas: emotional problems, behavioral problems, hyperactivity, relationship problems, and pro-social qualities.
The level of impulsivity assessed by the score of Impulsivity scale " UPPS Impulsive Behavior Scale ". | Day 0, month 3, month 6, month 12
  This scale (validated by Whiteside and Lynam, 2001) assesses impulsivity in adolescents, based on 4 components of impulsivity and 45 questions: urgency, lack of premeditation, lack of persistence and sensation seeking. If you put Absolutely, then it correspond to 1, if you just agree it correspond to 2, if you disagree it correspond to 3 and if you strongly disagree it is 4. Scoring is done so that a high score on a subscale corresponds to a higher level impulsivity => scores are obtained for Urgency, Lack of Premeditation, Lack of Perseverance, and Sensation Search.
Score of Self-esteem measurement scale (EMESA) to assess the adolescent's self-esteem. | Day 0, month 3, month 6, month 12
  This scale (validated by Kindelberger, Picherit, 2015) assesses adolescent self-esteem based on 5 areas of satisfaction: family, peers, schooling, professionalism and physical appearance.
Score of the DEP-ADO questionnaire to determine the addictions. | Day 0, month 3, month 6, month 12
  This grid is used to screen adolescents aged 11 to 17 for problematic alcohol and drug use. It is a questionnaire structured in 7 items, with a score that can range from 0 to greater than 17. A score of 0 to 8: no intervention, 9 to 16: intervention desirable, greater than 17: intervention necessary.
SDQ follow-up questionnaire | Month 3 and Month 6
  Questionnaire to determine whether the intervention solved or reduced the problems, whether the intervention was beneficial in making the problems more acceptable.
The level of therapeutic alliance assessed by the score of Therapeutic Alliance Questionnaire (CALPAS-T) | Month 3 and Month 6
  Evaluates the therapeutic alliance from the patient's point of view, according to four sub-scales: the patient's capacity for work, his commitment to therapy, the patient-therapist consensus on the work strategy, the therapist's involvement and understanding. The scale has 24 items, each rated from 0 to 7.
Score of Patient satisfaction Questionnaire (CSQ) to assess patient satisfaction. | Month 6
  This questionnaire collects the patient's opinion on its management.The questionnaire consists of 8 items, each rated from 1 to 4. Scores can range from 8 to 32. From 8 to 20, the level of satisfaction is low, from 21 to 26, the level is medium and from 27 to 32, the level of satisfaction is high.
Semi-structured interviews | Day 0, Month 3 and Month 6
  Done by assessors, other than those who will be performing the clinical assessment between T1 T2 and T3, using the RA interview guide to assess the subjective perception of the patient's mental suffering. Every professional on the team was trained in the methodology of the semi-directive interview.

CONTACTS AND LOCATIONS:
Locations (1):
- Etablissement Public de Santé de Ville-Evrard, Neuilly-sur-Marne, France

IPD SHARING:
Plan to Share IPD: No